CLINICAL TRIAL: NCT01160874
Title: Sleepiness and Performances Degradation in Adults Presenting an Attention-Deficit/ Hyperactivity Disorder (ADHD)
Brief Title: Sleepiness and Driving Performances in Adults With Attention-Deficit/ Hyperactivity Disorder (ADHD)
Acronym: SOMTDA/H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2009/17
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder / Hyperactivity (ADHD); Cognition; Sleepiness; Driving
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Sleepiness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TDA/H (Experimental)
  Interventions: Other: Polysomnography; Other: Maintenance Wakefulness Test; Behavioral: Neuropsychological evaluation; Other: Driving test on a simulator
- Sleep apnea patient (Other)
  Interventions: Other: Maintenance Wakefulness Test; Other: Driving test on a simulator
- Healthy volunteer (Other)
  Interventions: Other: Polysomnography; Other: Maintenance Wakefulness Test; Behavioral: Neuropsychological evaluation; Other: Driving test on a simulator

INTERVENTIONS:
Other: Polysomnography — Sleep study monitoring
  Arms: Healthy volunteer; TDA/H
Other: Maintenance Wakefulness Test — Sleep latency testing at 10 am, 12 am, 2 pm and 4 pm.
Behavioral: Neuropsychological evaluation — Neuropsychological evaluation for cognitive functions study
  Arms: Healthy volunteer; TDA/H
Other: Driving test on a simulator — Driving simulator test during wich a camera register different parameters as the position of the vehicle.

SUMMARY:
The Attention Deficit/ Hyperactivity Disorder (ADHD) is a developmental disorder which affects 3 to 5 % of school age children. This disorder persists in the adulthood for 60 % of subjects. Children with ADHD are sleepier during the day than normal children. However, there is no information concerning the diurnal sleepiness of adults with ADHD and the impact of this sleepiness on their driving capacity. The investigators postulate that the negative impact of ADHD is due to an awakening disorder which adds to the attentional disorder. The aim of this study is to estimate both the sleepiness by a Maintenance Wakefulness Test (MWT) and the capacity to drive in adults with ADHD.

DETAILED DESCRIPTION:
The main objective of this study is to estimate both the sleepiness by a Maintenance Wakefulness Test (MWT) and the capacity to drive in adults presenting an ADHD. Duration of participation for each patients will be 7 days. Four days after inclusion, patients will have to stop all psychostimulant treatment. Participants will then spend 24 hours (on days 6 and 7) at the "Groupe d'Etudes Neurophysiologie Pharmacologie Sommeil et Sommnolence"(GENPPHASS) in the "Centre Hospitalier Universitaire"(CHU) of Bordeaux. During this time, they will undergo complete polysomnography.The next day, they will perform a Maintenance Wakefulness Test (MWT). A neuropsychological evaluation of one hour will also be done. Finally, a driving test on a simulator will be performed.

Study significance: patients will benefit from an objective exploration of their sleep (with possibly, a sleep disorder discovery) and from a specific treatment. This study will demonstrate the necessity to investigate daytime function (sleepiness and performance) and the sleep quality of patients with ADHD. It will also demonstrate that part of the adults with ADHD handicap is based on an awakening disorder which adds to the attentional disorder.

ELIGIBILITY:
Inclusion Criteria:

Group for ADHD:

* Patients, male or female, aged 18 to 60 years
* Patients who met the criteria for current diagnosis of ADD / ADHD according to DSM IV-TR
* Patients who met the criteria for diagnosis in childhood ADD / ADHD, as assessed by the scale "Conners'Adult ADHD Diagnostic Interview for DSM-IV" (CCACID) (Conners, 1997)
* Patients with a total score ≥ 20 at the CAARS (hetero-questionnaire to 30 items) (Conners, 1997) with at least 6 items of inattention or hyperactivity subscale ≥ 2
* Patients deprived from all psychostimulants for 72 hours
* Having been schooled up to last year of middle school
* Having regular hours of life 3 days before entering the study
* Having a driver's license
* Registered Social Security
* Having given their written informed consent to participate in the study
* Consent free, informed and written, dated and signed by the patient and the investigator before any examination required by the research.

For the apneic group:

* Patients, male or female, aged 18 to 60 years
* Patients with apnea index of apnea / hypopnea> 10
* Having been schooled up to last year of middle school
* Having regular hours of life 3 days before entering the study
* Having a driver's license
* Registered Social Security
* Having given their written informed consent to participate in the study
* Consent free, informed and written, dated and signed by the patient and the investigator before any examination required by the research

For the control group:

* Participant male or female, aged 18 to 60 years
* Participant not symptomatic of ADHD (total score WURS less than 46 of the 25 questions about ADHD, and at least four more crosses in the boxes shaded the first 6 issues of ASRS)
* Participant with no complaints of sleep, or excessive daytime sleepiness (no item equal to 4 or 5 to BNSQ, except for items 16 and 17 (for snoring) and ESS total score below 11)
* Participant with an AHI <10 and MPS index <15 in ambulatory polygraph during the night of selection
* Participant with an AHI <10 and MPS Index <15 after overnight polysomnography in the laboratory prior to the day of testing
* Having been schooled until the third class,
* Having regular hours of life 3 days before entering the study,
* Having a driver's license,
* Registered Social Security,
* Having given their written informed consent to participate in the study
* Consent free, informed and written, dated and signed by the participant and the investigator before any examination required by the research.

Exclusion Criteria:

* Posted or Night worker,
* Any evolutionary neurological disorders (brain tumour, epilepsy, migraine, brain vascular accident, multiple sclerosis, myoclonus, chorea, neuropathy, muscular dystrophies, myotonic dystrophy),
* Psychiatric comorbidity: current major depressive episode, current hypo obsessive or obsessive episode, schizophrenia,
* Renal Disorders (renal insufficiency, nephrolithiases),
* Endocrine Pathologies (dysthyroid, diabetes),
* Drug addiction
* Alcoholic Dependence during the last 6 months,
* Dependence in the tetra-hydroxy-cannabinol
* Long-term Treatment by benzodiazépines
* Treatment by atomoxétine
* Persons placed under protection of justice

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Measurement of the average sleep latency during the Maintenance Wakefulness Test | Day 7

SECONDARY OUTCOMES:
The number of line crossing on the driving simulator test | Day 7
Standard deviation of the average position of the vehicle in the driving simulator test | Day 7
Score on Epworth Sleepiness scale | Day 7
Reaction time and the percentage of error in the cognitive tests | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Anouck AMESTOY, Dr, Principal Investigator — University Hospital Bordeaux (France)
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Charles Perrens, Bordeaux

REFERENCES:
- [Derived] Bioulac S, Chaufton C, Taillard J, Claret A, Sagaspe P, Fabrigoule C, Bouvard MP, Philip P. Excessive daytime sleepiness in adult patients with ADHD as measured by the Maintenance of Wakefulness Test, an electrophysiologic measure. J Clin Psychiatry. 2015 Jul;76(7):943-8. doi: 10.4088/JCP.14m09087. PMID 25610980